CLINICAL TRIAL: NCT07300449
Title: A Prospective Multicenter Clinical Study of the South China Collaborative Group Protocol for the Treatment of Hepatoblastoma in Children and Adolescents
Brief Title: A Prospective Multicenter Clinical Study of SCCG Protocol and ctDNA 5hmc in Predicting the Chemotherapy Sensitivity and Monitoring the Recurrence and Metastasis of Hepatoblastoma in Children and Adolescents
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Prof, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCG-HB
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hepatoblastoma
Keywords: hepatoblastoma
MeSH Terms: conditions — Hepatoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Very low-risk group (Experimental): The study used CHIC staging to stage hepatoblastoma
  Interventions: Drug: Very low-risk group; Other: 5hmc dynamic monitoring
- Arm 2: low risk group (Experimental): Patients received 2 to 4 courses of DDP monotherapy followed by elective surgery, then 2 additional courses of DDP monotherapy postoperatively, totaling 4 to 6 treatment cycles.
  Interventions: Drug: Low-risk group; Other: 5hmc dynamic monitoring
- Arm 3：intermediate risk group (Experimental): Treatment protocol randomization: Group A received SIOPEL-3 HR chemotherapy for 2-4 cycles followed by elective surgery, with continued chemotherapy for 6 additional cycles postoperatively.
  The patients in group B were given C5VD chemotherapy for 2-4 courses and then underwent elective operation.
  Interventions: Drug: Intermediate-risk group; Other: 5hmc dynamic monitoring
- Arm 4： High risk group (Experimental): Surgical resection after 3-5 courses of C-CD+ICE+solanifin chemotherapy
  Interventions: Drug: High-risk group; Other: 5hmc dynamic monitoring

INTERVENTIONS:
Drug: Very low-risk group — Very low-risk group: No chemotherapy after pure fetal type surgery, followed up and observed. Chemotherapy with other types of single-agent DDP regimens for 4 courses.
  Arms: Arm 1: Very low-risk group
Drug: Low-risk group — Low-risk group: 2 to 4 courses of DDP monotherapy chemotherapy, elective surgery, 2 courses of DDP monotherapy chemotherapy after surgery, totaling 4 to 6 courses.
  Arms: Arm 2: low risk group
Drug: Intermediate-risk group — Intermediate risk group: randomized treatment: group A SIOPEL - 3 HR solutions can be 2 ~ 4 course of chemotherapy, continue to A total of 6 course of chemotherapy after surgery. Group B C5VD solution after 2 ~ 4 course of chemotherapy, elective surgical procedures continue to a total of 6 course of chemotherapy after surgery.
  Arms: Arm 3：intermediate risk group
Drug: High-risk group — High-risk group：Chemotherapy with the C-CD+ICE+ sorafenib regimen for 3 to 5 courses was followed by elective surgery, with a total of 6 to 7 courses
  Arms: Arm 4： High risk group
Other: 5hmc dynamic monitoring — Peripheral blood was regularly drawn from patients in the very low-risk group, low-risk group, intermediate-risk group and high-risk group for 5hmc dynamic monitoring to evaluate its value in clinical efficacy and recurrence detection

SUMMARY:
Hepatoblastoma is the most common malignant liver tumor in infants and preschool children, comprising 65% of pediatric liver malignancies in those under 15, with its incidence on the rise in recent years [1]. Standard therapy combines surgical resection and chemotherapy: early-stage patients boast a survival rate over 90%, yet high-risk cases only reach around 40%, highlighting unmet treatment needs.

Notably, there is no universal definition for high-risk hepatoblastoma. The U.S. COG (AHEP0731) categorizes it as stage 4 disease, AFP <100ng/ml at diagnosis (any stage), or small cell undifferentiated histology; conversely, SIOP includes factors like major vascular invasion (inferior vena cava/portal vein), intra-abdominal extrahepatic spread, distant metastasis, AFP <100ng/ml, or tumor rupture, regardless of PRETEXT stage. To improve outcomes, international teams have tested intensified chemotherapy: Europe's SIOPEL reported that escalated cisplatin-doxorubicin regimens lifted high-risk patients' 3-year overall survival to over 80% [2], though with heightened toxicity. Similarly, Germany's IPA (ifosfamide-cisplatin-doxorubicin) and Japan's ITEC (ifosfamide-doxorubicin-carboplatin-VP-16) regimens delivered significant survival benefits but also amplified side effects [3,4].

Against this backdrop, the Guangdong Anti-Cancer Association's Pediatric Oncology Committee, led by Sun Yat-sen University Cancer Center and involving 15 hospitals, is launching a multicenter prospective trial to identify optimal chemotherapy regimens for Chinese hepatoblastoma children.

Parallelly, liquid biopsy has become an oncology research priority, offering four core advantages over tissue biopsy: non-invasiveness (peripheral blood sampling avoids tumor seeding), real-time genetic/progression monitoring (eliminating repeated invasive procedures), comprehensive molecular profiling (overcoming intratumoral heterogeneity), and high accuracy (capturing primary tumor-derived data). Given hepatoblastoma's propensity for early distant metastasis and 30-40% advanced-stage survival (with limited late-stage chemo efficacy), the Nano-5hmC-Seal cfDNA epigenetic profiling method holds promise as a novel biomarker for early diagnosis, treatment prediction, recurrence monitoring, and prognosis assessment in this disease.

DETAILED DESCRIPTION:
Sun Yat-sen University Cancer Center, the Guangdong Anti-Cancer Association's Pediatric Oncology Committee (15 participating hospitals) is launching a multicenter prospective trial to optimize chemotherapy for Chinese patients.

Liquid biopsy, with advantages of non-invasiveness, real-time monitoring, comprehensive profiling, and high accuracy, is an oncology priority. Given hepatoblastoma's early metastasis and poor advanced-stage outcomes (30-40% survival), Nano-5hmC-Seal cfDNA epigenetic profiling is a promising biomarker for diagnosis, treatment prediction, recurrence monitoring, and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary hepatoblastoma confirmed by pathology.

  * The age of the subjects was less than 18 years old. ③ Obtain the informed consent from the guardians and sign the informed consent form

Exclusion Criteria:

* Recurrent hepatoblastoma or other malignant tumor.

  * Age> 18 years old. ③ Patients with other tumors and received chemotherapy and abdominal radiotherapy.

    * Heart, brain and kidney failure patients.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | PFS is defined as the time interval from the start of treatment until the occurrence of disease progression or death of the patient from any cause, whichever happens first (up to 24 months）.
  progression of the disease or the death

SECONDARY OUTCOMES:
OS | The assessment of OS will be carried out over an estimated period of up to 24 months.
  Overall survival (OS) is defined as the time from the initiation of treatment with pucotenlimab in combination with theLenvatinib and Irinotecan regimen until the patient's death from any cause. Death is determined based on official medical records or other reliable documentation. The follow - up for OS will continue throughout this estimated assessment period.
Consistency | The assessment will be carried out over an estimated period of up to 24 months.
  The consistency of 5hmc dynamic monitoring in the evaluation of therapeutic effect and detection of tumor recurrence in hepatoblastoma in each risk group was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Junting Huang, Principal Investigator — SunYat Sen University Cancer Center; Huang, Study Director — SunYat Sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China